CLINICAL TRIAL: NCT04883229
Title: tDCS and Speech Therapy for Motor Speech Disorders Caused by FTLD Syndromes: a Feasibility Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The tDCS device that was going to be used for this study is no longer being made.
Sponsor: University of California, San Francisco (Other)
Collaborators: Halo Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: 18-26098
Record Dates: First submitted 2020-03-22; First posted 2021-05-12 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Nonfluent Aphasia, Progressive; Primary Progressive Nonfluent Aphasia; Primary Progressive Non Fluent Aphasia; Progressive Supranuclear Palsy; Corticobasal Degeneration; Behavioral Variant of Frontotemporal Dementia
Keywords: Motor Speech Disorders; Dysarthria; Apraxia of Speech
MeSH Terms: conditions — Primary Progressive Nonfluent Aphasia; Supranuclear Palsy, Progressive; Corticobasal Degeneration; Pick Disease of the Brain; Dysarthria; Apraxias | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- tDCS +speech therapy followed by sham tDCS + speech therapy (Experimental)
  Interventions: Device: Halo Neuroscience Neurostimulator
- sham tDCS +speech therapy followed by tDCS + speech therapy (Active Comparator)
  Interventions: Device: Halo Neuroscience Neurostimulator

INTERVENTIONS:
Device: Halo Neuroscience Neurostimulator — Experimental: Neurostimulation of 2 milliamps anodal (active) tDCS stimulation for 20 mins during 1 hour speech therapy sessions, 3 times a week for 8 weeks, plus daily homework. Then a washout period of no treatment, followed by a 8 weeks of sham tDCS treatment during 1 hour speech therapy sessions, 3 times a week for 8 weeks, plus daily homework.
  Active comparator: Experimental: Sham tDCS stimulation for 20 mins during 1 hour speech therapy sessions, 3 times a week for 8 weeks, plus daily homework. Then a washout period of no treatment, followed by a 8 weeks of neurostimulation of 2 milliamps anodal (active) sham tDCS treatment during 1 hour speech therapy sessions, 3 times a week for 8 weeks.
  Other Names: Speech therapy

SUMMARY:
The investigators will test the feasibility of using transcranial direct current stimulation (tDCS) and speech therapy to treat participants with motor speech disorders caused by Frontotemporal Lobar Degeneration Pathology including nonfluent variant Primary Progressive Aphasia, Progressive Supranuclear Palsy, Corticobasal Syndrome, or behavioral variant Frontotemporal Dementia.

The investigators will deliver transcranial direct current stimulation (tDCS) either in a clinic setting at the University of California San Francisco, or in patients' homes, via a consumer tDCS device and videoconferencing. Transcranial direct current stimulation (tDCS) is a neuromodulation technique that can enhance the benefits of speech therapy treatment. Participants will receive a dose of tDCS stimulation + speech therapy and a dose of sham tDCS + speech therapy in a randomized double blind crossover study performed either in the clinic or at home via videoconferencing. This study can be performed entirely remotely.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental Status Exam score > 10
* diagnosis of nfvPPA via Gorno-Tempini 2011 criteria, or a diagnosis of FTLD syndrome including progressive supranuclear palsy, corticobasal syndrome or behavioral variant frontotemporal dementia PLUS a motor speech disorder (apraxia of speech and/or dysarthria)
* able to give consent
* right-handed
* native English speaker
* having a caregiver who is also able to sign and understand the caregiver's consent form.

Exclusion Criteria: History of:

* stroke
* TBI
* brain cancer
* seizures
* craniotomy, skull surgery or fracture
* metallic implant in head
* pacemaker or cardioverter-defibrillator
* pregnancy.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in speech intelligibility | baseline and immediately after the first block of treatment
  Percent intelligible words, calculated by an SLP scoring each word spoken as intelligible or unintelligible, divided by total number of words spoken, during trained and untrained scripted speech.
Change in speech intelligibility | baseline and immediately after the second block of treatment
  Percent intelligible words, calculated by an SLP scoring each word spoken as intelligible or unintelligible, divided by total number of words spoken, during trained and untrained scripted speech.
Change in speech intelligibility | baseline and three months post treatment
  Percent intelligible words, calculated by an SLP scoring each word spoken as intelligible or unintelligible, divided by total number of words spoken, during trained and untrained scripted speech.

SECONDARY OUTCOMES:
Feasibility of remote use of device | Immediately after the second block of treatment
  Acceptability & ease of use of tDCS device from patient's homes. Measured via surveys designed by the investigators. Scores will range from 0 to 100. Higher scores will indicate better acceptability and ease of use.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Gorno Tempini, MD PhD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henry ML, Hubbard HI, Grasso SM, Mandelli ML, Wilson SM, Sathishkumar MT, Fridriksson J, Daigle W, Boxer AL, Miller BL, Gorno-Tempini ML. Retraining speech production and fluency in non-fluent/agrammatic primary progressive aphasia. Brain. 2018 Jun 1;141(6):1799-1814. doi: 10.1093/brain/awy101. PMID 29718131
- [Background] Tsapkini K, Frangakis C, Gomez Y, Davis C, Hillis AE. Augmentation of spelling therapy with transcranial direct current stimulation in primary progressive aphasia: Preliminary results and challenges. Aphasiology. 2014;28(8-9):1112-1130. doi: 10.1080/02687038.2014.930410. PMID 26097278
- [Background] Cotelli M, Manenti R, Ferrari C, Gobbi E, Macis A, Cappa SF. Effectiveness of language training and non-invasive brain stimulation on oral and written naming performance in Primary Progressive Aphasia: A meta-analysis and systematic review. Neurosci Biobehav Rev. 2020 Jan;108:498-525. doi: 10.1016/j.neubiorev.2019.12.003. Epub 2019 Dec 4. PMID 31811834
- [Background] Wang J, Wu D, Chen Y, Yuan Y, Zhang M. Effects of transcranial direct current stimulation on language improvement and cortical activation in nonfluent variant primary progressive aphasia. Neurosci Lett. 2013 Aug 9;549:29-33. doi: 10.1016/j.neulet.2013.06.019. Epub 2013 Jun 22. PMID 23800543
- [Background] Charvet L, Shaw M, Dobbs B, Frontario A, Sherman K, Bikson M, Datta A, Krupp L, Zeinapour E, Kasschau M. Remotely Supervised Transcranial Direct Current Stimulation Increases the Benefit of At-Home Cognitive Training in Multiple Sclerosis. Neuromodulation. 2018 Jun;21(4):383-389. doi: 10.1111/ner.12583. Epub 2017 Feb 22. PMID 28225155